CLINICAL TRIAL: NCT04811105
Title: OBLITERATION OF THE PERIANAL FISTULA TRACT BY STEAM ABLATION DEVICE IN THE TREATMENT OF PERIANAL FISTULA CAN BE USED AS A TREATMENT OPTION , A RAT STUDY
Brief Title: INVESTIGATION OF THE EFFICACY OF FISTULA OBLITERATION BY STEAM ABLATION IN PERİANAL FISTULAS
Acronym: STEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Asistant Dr , General Surgery , Principal Investigator,, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANIL ERGIN...
Record Dates: First submitted 2018-11-27; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Anal Fistula
Keywords: anal fistula; steam ablation; rat
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: 32 rats have 1 fistula tract 16 rats will treat with steam ablation 16 rats will be control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steam ablation (Active Comparator): The fistula tract which treated with steam ablation
  Interventions: Procedure: steam ablation
- control group (Active Comparator): The fistula tract which do not take any treatment
  Interventions: Procedure: steam ablation

INTERVENTIONS:
Procedure: steam ablation — 32 rats have 1 fistula tract .For 16 rats the investigator will use steam ablation to obliterate and 16 rats will be control group
  Other Names: perianal fistül treatment with steam ablation device

SUMMARY:
Perianal fistula(PF) is one of the most frequent disease in anorectal disease.The incidence of PF is 8,6 -10 / 100 000 . The first surgical treatment is defined by Hippocrates in PF .This surgical treatment which found by Hippocrates , involves seton insertion into the tract of fistula . Today most of surgeon still use the same technic but PF is really hard disease to treat. Recurrence rate of PF is really high and there are lots of complication about this disease. The most scary complication during the surgery or postoperatively is anal disfunction. ın PF surgical technics involves ;fistulectomy (coring out), lay open (fistulotomy), Ligation of Intersphincteric Fistula Tract, advancement flap and laser ablation of the fistula tract . The popularity of laser ablation of the fistula tract is increasing day by day.This surgical procedure is applied with the laser device which use in varicose vain ablation in vascular surgery.In this study the investigator are trying to find out the effect of steam ablation in PF on rats.

DETAILED DESCRIPTION:
Perianal fistula(PF) is one of the most frequent disease in anorectal disease..This surgical treatment which found by Hippocrates , involves seton insertion into the tract of fistula . Todaymost of surgeon still use the same technic but PF is really hard disease to treat. Recurrence rate of PF is really high and there are lots of complication about this disease.

The most scary complication during the surgery or postoperatively is anal disfunction. ın PF surgical technics involves ;fistulectomy (coring out), lay open (fistulotomy), Ligation of Intersphincteric Fistula Tract), advancement flap and laser ablation of the fistula tract . The popularity of laser ablation of the fistula tract is increasing day by day.This surgical procedure is applied with the laser device which use in varicose vain ablation in vascular surgery.In this study the investigator are trying to find out the effect of steam ablation in PF on rats.This new procedure has to be tried on rat firstly and the studies is very important which tried on rats.

Our research includes 32 rats and Firstly the investigator created perianal fistula tract with 2.0 silk suture material on 3 o'clock in perianal region.1 month will wait for the maturation of fistula tract. After that the suture materials removed from the fistula tract and one fistula tract will treat with steam ablation device (3 o'clock )in 16 rats and the other 16 rats will be the control group .1 month will be wait for the examination of treatment of fistula tract in steam ablation group.Evaluation of fistula tract will define with microscopic examination after the excision.End of the study the investigator will be find out the effect of steam ablation on perianal fistula .

ELIGIBILITY:
Inclusion Criteria:

* All rats which have iatrogenic perianal fistula tract.

Exclusion Criteria:

* Death of rat

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Perianal fistula is more frequent in male than woman nearly 8:1. So we have chosen the male rats
Enrollment: 16 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Effect of steam ablation treatment in perianal fistula in rats. | 7 weeks
  In the present study, we evaluated the effectiveness of steam ablation , associated or not to seton in the treatment of anal fistula surgically produced in rats. Although still very limited number of publications, the use of steam ablation in the treatment of anal fistula has shown promise, which was also observed in this study. There was a statistically significant difference when comparing the group treated with steam ablation and the control group. The previous seton placement not shown in this research any advantage, perhaps by allowing in some.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Medical School Experimental Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No